CLINICAL TRIAL: NCT05137418
Title: An Open-labelled, Bridging Phase Ⅲ Clinical Trial to Evaluate the Safety and Immunogenicity of COVID-19 Vaccine in Healthy Population Aged From 3 to 11 Years
Brief Title: Safety and Immunogenicity of COVID-19 Vaccine, Inactivated in Healthy Population Aged From 3 to 11 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCOV-3002-1
Record Dates: First submitted 2021-11-26; First posted 2021-11-30 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines; sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-5 years old age group (Experimental): 500 participants aged 3-5 years will receive two doses of COVID-19 vaccine,inactivated on day 0 and day 28.
  Interventions: Biological: COVID-19 Vaccine,Inactivated
- 6-11 years old age group (Experimental): 500 participants aged 6-11 years will receive two doses of COVID-19 vaccine,inactivated on day 0 and day 28.
  Interventions: Biological: COVID-19 Vaccine,Inactivated

INTERVENTIONS:
Biological: COVID-19 Vaccine,Inactivated — The COVID-19 vaccine,inactivated was manufactured by Sinovac Research& Development Co., Ltd..600SU Inactivated SARS-COV-2 virus in 0·5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac

SUMMARY:
This is an open-labelled, bridging phase Ⅲ clinical trial of COVID-19 Vaccine manufactured by Sinovac Research & Development Co., Ltd. The main purpose of this study is to evaluate the superiority of the COVID-19 Vaccine in healthy population aged from 3 to 11 years against that in adults aged 18-26 years.

DETAILED DESCRIPTION:
This study is a single-center, open-labelled, bridging phase Ⅲ clinical trial of COVID-19 Vaccine.The main purpose of this study is to evaluate the superiority of the COVID-19 Vaccine in healthy population aged from 3 to 11 years against that in adults aged 18-26 years.This study (PRO-nCOV-3002-1) will be used as a sub-trial of the Phase Ⅲ global multi-center clinical trial in children and adolescents(PRO-nCOV-3002) to provide safety and immunogenicity data.A total of 1000 healthy children aged 3-11 years will be enrolled ,including 500 children aged 3-5 years and 500 children aged 6-11 years.All subjects will receive 2 doses of experimental vaccine (600SU) with an interval of 28 days,and adverse reactions/events will be collected from all subjects after each dose and SAE and AESI monitoring will be completed from the beginning of vaccination to 6 and 12 months after full vaccination to evaluate the safety of the vaccine.About 3.0-3.5ml of venous blood will be collected from all subjects before immunization, 28 days after the whole immunization, 6 months after the whole immunization and 12 months after the whole immunization. Neutralizing antibody and S antibody will be detected to evaluate the immunogenicity and immune persistence of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged 3-11 years;
* The participants and/or their guardians are able to understand and sign the informed consent voluntarily (in accordance with the local regulations)(For subjects aged 3-7years ,guardians need to sign the informed consent form,for subjects aged 8-17 years, both subjects and guardians need to sign the informed consent form);
* Able to comply with study procedures based on the assessment of the Investigator
* Must be willing to provide verifiable identification (in accordance with the local regulations), has means to be contacted and to contact the investigator during the study.

Exclusion Criteria:

* History of SARS-CoV-2 infection;
* Close contact with a confirmed COVID-19 within 14 days prior to randomization;
* Prior administration of an investigational coronavirus vaccine or current/ planned simultaneous participation in another interventional study to prevent or treat COVID-19;
* Allergy to vaccines or vaccine/placebo ingredients, and serious adverse reactions to vaccines, such as urticaria, dyspnea, angioneuroedema;
* Personal or first-grade relative (siblings) history of multisystem inflammatory disease in children (MIS-C);
* Significant chronic illnesses that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion (may include, but are not limited to cardiovascular disease, liver or kidney disorders, respiratory illnesses);
* Significant chronic central nervous system diseases or neuromuscular disorders, psychosis or severe cognitive behavioral disorder, in the opinion of the investigator, including epilepsy, autism spectrum disorder, intellectual disabilities (excluding Down Syndrome);
* Acute central nervous system diseases such as encephalitis/myelitis, acute disseminating encephalomyelitis, and related disorders;
* History of autoimmune and/or haematological diseases (including but not limited to systemic lupus erythematosus, thyroidectomy, autoimmune thyroid disease, any form of malignant tumor, asplenia, functional asplenia, or splenectomy resulting from any condition); well controlled type I diabetes mellitus is allowed;
* History of bleeding disorders (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture;
* Immunosuppressive therapy (systemic corticoid therapy, e.g. prednisone

  ≥2 mg/Kg/d or ≥20 mg/day for >14 days), cytotoxic therapy (antineoplastic chemotherapy, radiation therapy), (excluding topical or aerosol corticosteroid therapy) in the past 6 months;
* Receipt of blood products or immunoglobulins in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute exacerbation or presentation of stable chronic diseases (including but not limited to asthma, migraine, gastrointestinal disorder, etc;
* Acute febrile illness with oral temperature >37.7°C ,enrollment could be considered if the fever is absent for 72 hours;
* Any confirmed or suspected human immunodeficiency virus (HIV) infection;
* Children in care or under a court order;
* According to the investigator's judgment, the subject has any other factors that might interfere with the results of the clinical trial or pose additional risk to the subject due to participation in the study.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2021-11-27 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index-the GMT of neutralizing antibodies | 28 days after the second vaccination
  The GMT of neutralizing antibodies 28 days after the second vaccination.

SECONDARY OUTCOMES:
Immunogenicity index-the seroconversion rate of neutralizing antibodies | 28 days after the second vaccination
  The seroconversion rate of neutralizing antibodies 28 days after the second vaccination
Immunogenicity index-the seropositive rate of neutralizing antibodies 28 days after the second vaccination | 28 days after the second vaccination
  The seropositive rate of neutralizing antibodies 28 days after the second vaccination
Immunogenicity index-GMI of neutralizing antibodies | 28 days after the second vaccination
  GMI of neutralizing antibodies 28 days after the second vaccination
Immunogenicity index-The seroconversion rate of the S antibody to SARS-CoV-2 | 28 days after the second vaccination
  The seroconversion rate of the S antibody to SARS-CoV-2 28 days after the second vaccination
Immunogenicity index-The seropositivity rate of the S antibody to SARS-CoV-2 | 28 days after the second vaccination
  The seropositivity rate of the S antibody to SARS-CoV-2 28 days after the second vaccination
Immunogenicity index-GMC of the S antibody to SARS-CoV-2 | 28 days after the second vaccination
  GMC of the S antibody to SARS-CoV-2 28 days after the second vaccination
Immunogenicity index-GMI of the S antibody to SARS-CoV-2 | 28 days after the second vaccination
  GMI of the S antibody to SARS-CoV-2 28 days after the second vaccination
Immunogenicity index-The seropositive rate of neutralizing antibodies | 6 months/12 months days after the second vaccination
  The seropositive rate of neutralizing antibodies 6 months/12 months days after the second vaccination
Immunogenicity index-GMT of neutralizing antibodies | 6 months/12 months days after the second vaccination
  GMT of neutralizing antibodies 6 months/12 months days after the second vaccination
Immunogenicity index-The seropositivity rate of the S antibody to SARS-CoV-2 | 6 months/12 months days after the second vaccination
  The seropositivity rate of the S antibody to SARS-CoV-2 6 months/12 months days after the second vaccination
Immunogenicity index-GMC of the S antibody to SARS-CoV-2 | 6 months/12 months days after the second vaccination
  GMC of the S antibody to SARS-CoV-2 6 months/12 months days after the second vaccination
Safety index-Incidence rate of adverse reactions | From the beginning of the vaccination to 28 days after the second dose vaccination
  Incidence rate of adverse reactions occured from the beginning of the vaccination to 28 days after the second dose vaccination
Safety index-Incidence rate of SAEs | From the beginning of the vaccination to 6 months after the second dose vaccination
  Incidence rate of SAEs from the beginning of the vaccination to 6 months after the second dose vaccination.
Safety index-Incidence rate of AESIs | From the beginning of the vaccination to 6 months after the second dose vaccination
  Incidence rate of AESIs from the beginning of the vaccination to 6 months after the second dose vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Pan, Master, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (1):
- Sheyang County Center for Disease Control and Prevention, Yancheng, Jiangsu, China